CLINICAL TRIAL: NCT00199030
Title: German Multicenter Phase II Trial to Study Effectivity and Feasibility of Alemtuzumab (MabCampath®) in T-ALL and T-Lymphoblastic Lymphomas With Minimal Residual Disease (MRD), in Refractory Relapse or in Primary Failure
Brief Title: Treatment of Relapsed T-cell Acute Lymphoblastic Leukemia or T-lymphoblastic Lymphoma With MabCampath
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Head of GMALL, Goethe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMALL07
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Adult Acute Lymphocytic Leukemia T-cell; Lymphoma, Lymphoblastic
Keywords: Relapse; T-ALL; T-LBL; MabCampath; Minimal residual disease; Lymphoma, lymphoblastic, T-cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual; Lymphoma | interventions — Alemtuzumab; Cladribine

STUDY DESIGN:
Intervention Model Description: 2 arms; Allocation by stratification
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): In Arm A, patients with refractory relapse receive a 2 week treatment with MabCampath followed by remission evaluation. In case of insufficient response, treatment with cladribine is added.
  Interventions: Drug: Alemtuzumab (MabCampath); Drug: Cladribine
- Arm B (Experimental): In Arm B, patients with molecular relapse (minimal residual disease) receive a 4 week treatment with MabCampath followed by remission evaluation.
  Interventions: Drug: Alemtuzumab (MabCampath)

INTERVENTIONS:
Drug: Alemtuzumab (MabCampath)
Drug: Cladribine
  Arms: Arm A

SUMMARY:
This study tests the effectivity and tolerability of treatment with alemtuzumab (MabCampath) in patients with relapsed or refractory T-cell acute lymphoblastic leukemia (T-ALL) or T-lymphoblastic lymphoma. In Arm A, patients with refractory relapse receive a 2 week treatment with MabCampath followed by remission evaluation. In case of insufficient response, treatment with cladribine is added. In Arm B, patients with molecular relapse (minimal residual disease) receive a 4 week treatment with MabCampath followed by remission evaluation. In both arms, treatment is continued in case of response for up to two months.

ELIGIBILITY:
Inclusion Criteria:

Both Arms:

* T-ALL or T-lymphoblastic lymphoma
* CD52-expression > 20%
* Aged >= 18 years
* ECOG/World Health Organization (WHO) performance status 0-2
* Life expectancy of > 2 months
* Contraception during, and for at least 6 months after, therapy
* At least a 2 week interval to the last cycle of chemotherapy (decision in individual cases if rapid progression)
* No persistent toxicity from earlier cycles
* Written informed consent

Arm 1:

* Evidence of MRD > 10(-4) with confirmation beyond week 16 in the GMALL-Study 07/2003

Arm 2:

* Relapse with failure to at least one salvage therapy or primary failure after induction therapy and at least one salvage therapy

Exclusion Criteria:

* Substantial restrictions of heart, lung, liver, or kidney function
* Active infection, HIV seropositivity or cytomegalovirus (CMV) viraemia
* Pretreatment with MabCampath®
* Known anaphylaxis to humanised antibodies
* Permanent systemic therapy with corticosteroids
* Central nervous system (CNS) involvement
* Extramedullary bulky disease
* Active secondary malignancies
* Pregnancy or nursing
* Mental disease or circumstances that prohibit compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Arm A: rate of molecular remissions (MRD < 10(-4), toxicity according to CTC, remission duration/survival, feasibility of s.c. dose escalation and long term therapy, mortality | after 1 cycle - approximately 3 weeks
Arm B: response (CR/PR/MR), toxicity according to CTC, SCT rate, remission duration/survival, feasibility of i.v. dose escalation/long term therapy, mortality | after 1 Cycle - approximately 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Study Chair — University Hospital Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany